CLINICAL TRIAL: NCT04951011
Title: Different Treatment Options for Tubal Ectopic Pregnancy:- A Systmatic Review
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelhameed Mohamed, resident doctor at obstitrics and gyncology department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-06-05
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Woman With Tubal Ectopic Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum beta HCG — Raising numbers of S BHCG or decreasing with different management of tubal Ectopic Pregnancy

SUMMARY:
Ectopic pregnancy is an early pregnancy complication in which a fertilized ovum implant outside the uterine cavity. Implantation may occur anywhere along the reproductive tract with the most common implantation site being the fallopian tube. The incidence of ectopic pregnancy is 1% of pregnant women, and may seriously compromise women's health and future fertility.

Currently, ectopic pregnancy can be often diagnosed before the woman's condition has deteriorated, which has altered the former clinical picture of a lifethreatening disease into a more benign condition in frequently asymptomatic women.

ELIGIBILITY:
Inclusion criteria:

* RCTs and observational studies
* All types of ectopic pregnancies.
* All types of treatments and medications for ectopic pregnancies.
* The long-term survival of patients with or without complications.
* Successful pregnancy and birth.

Exclusion criteria:

* Articles of failed treatments of ectopic pregnancies.
* Articles with over all P value > 0.05.
* Articles for which the full text is not available in English.

Ages: 15 Years to 40 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Sample size: All articles fulfilling the inclusion criteria within the last five years.
  Study tools: Primary data will be re-analyzed statistically and processed data to be compared. Secondary data will be analyzed for correlation between the type of anastomosis (hand sewing vs. staplers) and between measurements outcome (leakage and, stricture and fistula formation).
  • Study procedure: The study will start by searching articles using the key words and then downloading papers that fulfill the inclusion criteria and excluding papers with exclusion criteria. These papers will be examined by the supervisors to make sure of finding the appropriate source of data and then I will start working with the statistical supervisor and put data on R-based software for meta-analysis and start conducting the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal and Transvaginal Ultrasound: | 6 Monthes
  To detect the appearance of any mass at the adenexa,or intrauterine gestational sac in case of heterotopic pregnancy or misdiagnosis of ectopic pregnancy.
  To detect, if there's collection at the pelvis or freely at the abdomen in the case of disturbed ectopic pregnancy.
S.bHCG: | 6 Monthes
  in cases of expectant management,and medical treatment to detect level of S.bHCG after administration of methotrexate to decide to continue with medical treatment and give another doses or failure of this line and decide another line of management.
  Also,at the expectant management to close follow up the patient.
Diagnostic laparoscopy | 6 Monthes
  In cases of early,undisturbed ectopic pregnancy and may use also,for therapy Laparoscopic salpingostomy and/or salpingectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag, Akhmīm, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Barnhart KT. Clinical practice. Ectopic pregnancy. N Engl J Med. 2009 Jul 23;361(4):379-87. doi: 10.1056/NEJMcp0810384. No abstract available. PMID 19625718
- [Background] Bagshawe KD, Dent J, Newlands ES, Begent RH, Rustin GJ. The role of low-dose methotrexate and folinic acid in gestational trophoblastic tumours (GTT). Br J Obstet Gynaecol. 1989 Jul;96(7):795-802. doi: 10.1111/j.1471-0528.1989.tb03318.x. PMID 2548568
- [Background] Elson J, Tailor A, Banerjee S, Salim R, Hillaby K, Jurkovic D. Expectant management of tubal ectopic pregnancy: prediction of successful outcome using decision tree analysis. Ultrasound Obstet Gynecol. 2004 Jun;23(6):552-6. doi: 10.1002/uog.1061. PMID 15170794